CLINICAL TRIAL: NCT04959279
Title: A Pilot Randomized Controlled Trial of ED-TREAT (Early Detection and Treatment to Reduce Events With Agitation Tool) Compared to Usual Care
Brief Title: ED-TREAT (Early Detection and Treatment to Reduce Events With Agitation Tool) Compared to Usual Care
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is in process of transferring to a new institution
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000030906; K23MH126366-01A1 (NIH)
Record Dates: First submitted 2021-06-30; First posted 2021-07-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Psychomotor Agitation; Behavioral Disorder
MeSH Terms: conditions — Psychomotor Agitation; Mental Disorders

STUDY DESIGN:
Intervention Model Description: 2:1 randomization and also recruit a higher proportion of high-risk patients in each arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ED-TREAT (Experimental): EHR-embedded clinical decision support (CDS) tool designed to overcome the challenges to risk assessment and suggest pre-emptive use of behavioral techniques in the emergency setting.
  Interventions: Other: ED-TREAT
- Usual Care (No Intervention)

INTERVENTIONS:
Other: ED-TREAT — Patients will be assessed and treated based on a clinical decision support system.
  Arms: ED-TREAT

SUMMARY:
The purpose of this study is to conduct a a pilot trial that tests the acceptability, fidelity, and feasibility of ED-TREAT.

DETAILED DESCRIPTION:
This study will be a pilot RCT that compares ED-TREAT to usual care. The scientific premise of the proposed project is that an innovative EHR-embedded clinical decision support (CDS) tool can overcome the challenges to risk assessment and suggest pre-emptive use of behavioral techniques in the emergency setting. This would help clinicians appropriately invest resources to improve the quality of care for at-risk patients regardless of ultimate medical or psychiatric diagnoses and prevent agitation from occurring.

This pilot trial will (1) test the integrity of the study protocol in preparation for a future full-scale RCT, (2) evaluate randomization protocols, (3) estimate rates of recruitment and retention, (4) assess acceptability and fidelity of the intervention, and (5) determine if the proposed effect size is reasonable.

This registered study is actually the third aim of a larger study where the tool will be developed and assessed using observational data and input from a steering committee in aims 1 and 2 prior to pilot testing.

ELIGIBILITY:
Inclusion Criteria:

1. adult (age≥18) patients presenting to the YNHH ED during the pilot trial period
2. deemed to have a mild-moderate or high risk of agitation as determined by ED-TREAT
3. do not require physical restraint orders <30 minutes of arrival
4. with a score of "4" (quiet and awake; normal level of activity) on the Behavioral Activity Rating Scale
5. have comfort with conversational English
6. able to provide verbal consent.

Exclusion Criteria:

1. Presence of a restraint order <30 minutes of arrival and presence of a non-violent physical restraint order where indications are not due to agitation (e.g., for protecting intubation or life-preserving equipment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of visits adherent to protocol | 12 months
  Proportion of visits in the intervention arm that are adherent to >95% of the observational workflow checklist (primary outcome of fidelity)

SECONDARY OUTCOMES:
System usability scale | Baseline, 15 hours
  Acceptability will be measured using a scale the System Usability Scale. The System Usability Scale is a widely used and effective survey composed of ten statements assessed on a 5-point Likert scale, with inter-item correlations of 0.69-0.75 and a reliability coefficient α of 0.91. The scale provides continuous data from 0-100 with scores >85 as indicative of excellent usability, and will be described using mean and standard deviation. The study will consider ED-TREAT to be acceptable if at least 90% of each clinician group give ratings >85.

CONTACTS AND LOCATIONS:
Overall Officials: Ambrose H. Wong, (203) 737-2489, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong AH, Nath B, Shah D, Kumar A, Brinker M, Faustino IV, Boyce M, Dziura JD, Heckmann R, Yonkers KA, Bernstein SL, Adapa K, Taylor RA, Ovchinnikova P, McCall T, Melnick ER. Formative evaluation of an emergency department clinical decision support system for agitation symptoms: a study protocol. BMJ Open. 2024 Feb 19;14(2):e082834. doi: 10.1136/bmjopen-2023-082834. PMID 38373857